CLINICAL TRIAL: NCT05733897
Title: Using Hydroxychloroquine to Treat Nonalcoholic Steatohepatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Sponsor
Other Study IDs: 202206002RINB
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic Steatohepatitis; Hydroxychloroquine; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Hydroxychloroquine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: hydroxychloroquine — Using hydroxychloroquine to treat nonalcoholic steatohepatitis
  Other Names: Plaquenil®

SUMMARY:
Nonalcoholic steatohepatitis (NASH) is a serious type of nonalcoholic fatty liver disease (NAFLD), which is characterized by lobular inflammation and apoptosis resulting from hepatic steatosis in the absence of excessive alcohol consumption. If NASH are not controlled well, it will advance to liver fibrosis, cirrhosis, and even hepatocellular carcinoma. However, there is no approved treatments currently.

The investigators aim to clarify whether hydroxychloroquine relieves nonalcoholic steatohepatitis by reviewing medical records from our out-patient-clinic patients who accept the treatment of hydroxychloroquine (Plaquenil®).

DETAILED DESCRIPTION:
Nonalcoholic steatohepatitis (NASH) is a serious type of nonalcoholic fatty liver disease(NAFLD), which is characterized by lobular inflammation and apoptosis resulting from hepatic steatosis in the absence of excessive alcohol consumption. If NASH are not controlled well, it will advance to liver fibrosis, cirrhosis, and even hepatocellular carcinoma. However, there is no approved treatments currently.

According to guidance of American Association for the Study of Liver Diseases (AASLD) and a few studies, vitamin E and pioglitazone are two potential pharmacologic therapies for NASH. They have some therapeutic effects; however, they also have some safety concerns. Therefore, those two drugs have not been wildly used in clinical practices. In addition to vitamin E and pioglitazone, many drugs are being tested in clinical trials. However, promising results have not been revealed yet.

Recent clinical and experimental data suggested that hydroxychloroquine (HCQ) might improve metabolic profiles in patients or animals with obesity-related metabolic disorders. HCQ might also relieve liver inflammation in experimental animals with steatohepatitis. As an inhibitor of endocytosis and autophagy with therapeutic effects in autoimmune disorders, it is reasonable to speculate that HCQ might also relieve liver inflammation in patients with steatohepatitis. Therefore, HCQ has been anecdotally prescribed to patients with steatohepatitis in our clinic. Excitingly, almost all those with HCQ treatment had immediate reduction of their liver enzyme levels, indicating instant relief of their steatohepatitis. Effects of HCQ were similar in those with negative anti-nuclear antibody (ANA) compared to those with weakly positive ANA, suggesting that those are specific steatohepatitis-targeting rather than autoimmune-targeting effects from HCQ.

Thus, the investigators aim to clarify whether HCQ relieves nonalcoholic steatohepatitis by reviewing medical records from our out-patient-clinic patients who accept the treatment of hydroxychloroquine (Plaquenil®).

ELIGIBILITY:
screen out our targeted group：patients with nonalcoholic steatohepatitis

1. The investigators have made a request to Information Technology Office of National Taiwan University Hospital, and this request is about the list of our out-patient-clinic patients who accept the treatment of hydroxychloroquine.
2. Collect and review the medical records, ultrasound and blood tests of patients in the abovementioned list and screen out those with nonalcoholic steatohepatitis based on the following criteria.

Inclusion criteria： Our patients who taking hydroxychloroquine and match the following criteria

A. Patients with fatty liver, based on the abdominal ultrasound report of which the date is the closest to the initial date of using HCQ.

B. Alanine aminotransferase (ALT) level of 2.5 and 0.5 month prior to hydroxychloroquine treatment > 41 U/L

C. With ALT result which is tested in 3 months after using HCQ.

D. The initial date of taking HCQ is prior to September, 26, 2022, which is the date we got the list from Information Technology Office of National Taiwan University Hospital.

Exclusion criteria： Our exclusion criteria can be separated into loose exclusion criteria and strict exclusion criteria.

Loose exclusion criteria：patients who match the following criteria will be excluded from the above group.

A. Diseases of the biliary tract：the abdominal ultrasound report indicated the patient with stones in the biliary tract, or the patient with jaundice or his total bilirubin > 2.0 mg/dl

B. Viral hepatitis： Hepatitis B Virus (HBV) Viral Load + or Hepatitis C Virus (HCV) Viral Load +

C. Alcoholic steatohepatitis： History of drinking alcohol or aspartate aminotransferase /alanine aminotransferase (AST/ALT) > 1.5 and γ-glutamyltransferase (GGT) > two times of normal levels (2X)

D. Autoimmune hepatitis： anti-nuclear antibody (ANA)1:80+ (above) or mitochondrial antibody (AMA) + or liver kidney microsome antibody (anti-LKM) + or smooth muscle antibody (anti-SMA) +

E. Wilson's disease：ceruloplasmin < 20 mg/dl

Strict exclusion criteria：patients who had ever had viral hepatitis or was being infected by virus (HBV, HCV infection：hepatitis B surface antigen positive (HBsAg+) or hepatitis B core antibody positive (HBc stands for hepatitis B core antigen, anti-HBc+ stands for hepatitis B core antibody) or anti-HCV Ab+) will be further excluded from the above group.

The definition of months：used in the criteria evaluation and the data analysis

Before patients used HCQ：

negative 0.5 month：During the periods from one month prior to the date of initial use of HCQ to that date, we define the date which is the closest to 0.5 month as -0.5 month.

negative 2.5 months：During the periods from four months to one month prior to the date of initial use of HCQ, we define the date which is the closest to 2.5 months as -2.5 months.

negative 5.5 months：During the periods from seven months to four months prior to the date of initial use of HCQ, we define the date which is the closest to 5.5 months as -5.5 months.

After patients used HCQ： 0.75 months：During the periods that patients used HCQ for 0-1.5 months, we define the date which is the closest to 0.75 months as 0.75 months.

3 months：During the periods that patients used HCQ for 1.5-4.5 months, we define the date which is the closest to 3 months as 3 months.

6 months：During the periods that patients used HCQ for 4.5-7.5 months, we define the date which is the closest to 6 months as 6 months.

9 months：During the periods that patients used HCQ for 7.5-10.5 months, we define the date which is the closest to 9 months as 9 months.

12 months：During the periods that patients used HCQ for 10.5-13.5 months, we define the date which is the closest to 9 months as 12 months.

Then, in addition to the above-mentioned criteria, we will record the following two things separately.

The first one is hemochromatosis. Hemochromatosis may also cause hepatitis, but the prevalence of this disease in Taiwan is very low. Thus, we do not list hemochromatosis in the exclusion criteria.

The second one is drug-induced hepatitis. We do not list suspected drug-induced hepatitis in the exclusion criteria since drug-induced hepatitis may not be accurately confirmed based on our current medical records. However, if we find patients using drugs which may be related to hepatitis, we will record their information separately, including the duration of using these drugs and the ALT levels after stopping using it.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study population are collected from our out-patient-clinic patients who accept the treatment of hydroxychloroquine.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
To observe whether patients' alanine aminotransferase (ALT) levels were significantly decreased after using hydroxychloroquine (by statistically analyzing patients' ALT levels before and after using HCQ) | during the period of one year after taking hydroxychloroquine
  Comparing patients' alanine aminotransferase (ALT) levels before using hydroxychloroquine with those after using hydroxychloroquine, to observe whether ALT levels were significantly decreased (by statistically analyzing patients' ALT levels before and after using HCQ).

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Jui Huang, Master, Study Director — Graduate Institute of Pharmacology, College of Medicine, National Taiwan University; Feng-Chiao Tsai, Doctor, Principal Investigator — Graduate Institute of Pharmacology, College of Medicine, National Taiwan University
Locations (2):
- Taiwan (2):
  - Graduate Institute of Pharmacology, College of Medicine, National Taiwan University, Taipei
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Background] Pouwels S, Sakran N, Graham Y, Leal A, Pintar T, Yang W, Kassir R, Singhal R, Mahawar K, Ramnarain D. Non-alcoholic fatty liver disease (NAFLD): a review of pathophysiology, clinical management and effects of weight loss. BMC Endocr Disord. 2022 Mar 14;22(1):63. doi: 10.1186/s12902-022-00980-1. PMID 35287643
- [Background] Niture S, Lin M, Rios-Colon L, Qi Q, Moore JT, Kumar D. Emerging Roles of Impaired Autophagy in Fatty Liver Disease and Hepatocellular Carcinoma. Int J Hepatol. 2021 Apr 22;2021:6675762. doi: 10.1155/2021/6675762. eCollection 2021. PMID 33976943
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] Wong SK. Repurposing New Use for Old Drug Chloroquine against Metabolic Syndrome: A Review on Animal and Human Evidence. Int J Med Sci. 2021 May 13;18(12):2673-2688. doi: 10.7150/ijms.58147. eCollection 2021. PMID 34104100
- [Background] Qiao X, Zhou ZC, Niu R, Su YT, Sun Y, Liu HL, Teng JL, Ye JN, Shi H, Yang CD, Cheng XB. Hydroxychloroquine Improves Obesity-Associated Insulin Resistance and Hepatic Steatosis by Regulating Lipid Metabolism. Front Pharmacol. 2019 Aug 2;10:855. doi: 10.3389/fphar.2019.00855. eCollection 2019. PMID 31427967
- [Background] Schrezenmeier E, Dorner T. Mechanisms of action of hydroxychloroquine and chloroquine: implications for rheumatology. Nat Rev Rheumatol. 2020 Mar;16(3):155-166. doi: 10.1038/s41584-020-0372-x. Epub 2020 Feb 7. PMID 32034323